CLINICAL TRIAL: NCT05173324
Title: Integration of HPV Vaccination and HPV-based Cervical Screening in Young Adult WLWH Into ARV Clinics to Speed the Pathway Towards Cervical Cancer Elimination: the H2VICTORY Trial
Brief Title: Integration of HPV Vaccination and HPV-based Cervical Screening Into ARV Clinics: the H2VICTORY Trial
Acronym: H2VICTORY
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: University of New Mexico (Other); University of Stellenbosch (Other); University of KwaZulu (Other); Coptic Hope Center (Unknown); Emory University (Other); Ministry of Health, Swaziland (Other Government); Baylor College of Medicine Children's Foundation (Unknown); Sefako Makgatho Health Sciences University (Other); Aga Khan University (Other); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PP202111-31
Record Dates: First submitted 2021-12-15; First posted 2021-12-29 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: HPV Infection
Keywords: HPV vaccination; HPV-based cervical screening; HIV infection; Cervical ablative treatment; Antiretroviral clinics; Implementation research; Hybrid effectiveness-implementation trials
MeSH Terms: conditions — Papillomavirus Infections; HIV Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- 3-doses HPV vaccination (Experimental): Participants will receive three doses of HPV vaccine at 0, 2, and 6 months
  Interventions: Biological: HPV vaccine; Diagnostic Test: HPV testing
- 1-dose HPV vaccination (Experimental): Participants will receive HPV vaccine at entry, and placebo (HAV vaccine) at 2 and 6 months
  Interventions: Biological: HPV vaccine; Diagnostic Test: HPV testing; Biological: HAV vaccine
- Placebo (Placebo Comparator): Participants will receive Hepatitis A (HAV) vaccine at 0, 2, and 6 months
  Interventions: Diagnostic Test: HPV testing; Biological: HAV vaccine

INTERVENTIONS:
Biological: HPV vaccine — Licensed HPV vaccines (bivalent, quadrivalent, or nonvalent) available in the country of the study site
  Arms: 1-dose HPV vaccination; 3-doses HPV vaccination
Diagnostic Test: HPV testing — HPV testing with partial genotyping of HPV16/18 (and/or 45) to be used as a primary cervical screening test for all participants regardless of the study arm
Biological: HAV vaccine — Hepatitis A virus (HAV) vaccine to be offered as a placebo
  Arms: 1-dose HPV vaccination; Placebo

SUMMARY:
A 3-dose HPV vaccination scheme has shown to be safe and immunogenic in people living with HIV (PLWH), although evidence on 1-dose, which is important to improve coverage, is scarce. Available HPV vaccines only prevent new infections. Since a large fraction of WLWH is already infected with HPV (>50%), vaccines' efficacy to prevent HPV infections (and therefore cervical disease) in this population is limited. Current WHO cervical cancer screening guidelines recommend treatment of the transformation zone (TZ) of WLWH who harbor HPV infections either at initial screening or one year later. Therefore, HPV vaccination at the time of the screening may improve vaccines efficacy conferring protection to newly growing cells of the treated TZ against HPV infections/re-infections. Consequently, a dual-intervention of HPV vaccination and HPV-based cervical screening in WLWH may alleviate the burden of HPV-related disease by improving HPV vaccination efficacy while extending cervical screening intervals. Nevertheless, implementing the dual-intervention may be challenging particularly in some contexts without well-established cervical cancer screening such as sub-Saharan African (SSA) countries. However, in these countries, at least 60% of PLWH regularly attend ARV clinics to be monitored and receive ARV treatment (cART). Therefore, integrating the dual-intervention into ARV clinics seems to be an efficient approach to reduce loss to follow-up while improving overall coverages of HPV vaccination and cervical screening. Such integration may also facilitate the implementation of a platform for the delivery of other HPV-related preventive measures such as HPV therapeutic vaccines.

Nevertheless, little is known about the efficacy of HPV vaccination in WLWH to prevent HPV infections and HPV-related diseases, especially in young adults. Moreover, evidence on how best to conduct cervical cancer prevention, particularly recently released WHO guidelines, through ARV clinics is limited. Therefore, IARC/WHO in collaboration with HRP/WHO and colleagues in SSA proposes to conduct a hybrid effectiveness-implementation trial (H2VICTORY) to evaluate the effectiveness of the dual-intervention of HPV vaccination and HPV-based cervical screening to reduce HPV infections (and therefore, the risk of cervical cancer) in WLWH aged 25-35 years while conducting implementation research to identify facilitators and barriers for adoption and sustainability of proven evidence-based cervical cancer prevention approaches integrated into ARV clinics across sub-Saharan Africa.

DETAILED DESCRIPTION:
An effectiveness-implementation hybrid study is proposed to evaluate the effectiveness of a dual intervention of HPV vaccination and HPV-triage-and-treat to reduce the risk of cervical cancer and to study its integration into ARV clinics. The overarching hypothesis will be that offering the dual intervention of HPV vaccination and HPV-triage-treat in young WLWH will catalyze the preventive effect of both evidence-based interventions as: (i) the HPV vaccination efficacy will be improved when applied after HPV infections are (progressively) removed by treatment of the TZ (enrolment, 12 months, both) as the vaccine will confer protection from new infections to new TZ growing cells; and (ii) the reduction of new HPV infections may allow extension of HPV-triage-treat intervals, contributing to feasible scale-up of comprehensive cervical cancer preventive care to WLWH attending ARV clinics. The H2VICTORY specific aims are:

1. To assess the readiness ARV clinics in sub-Saharan African countries to inform contextually relevant strategies to de-implement current interventions (i.e. Pap, VIA) and implement and integrate the dual-intervention of HPV vaccination and HPV-based cervical screening and treatment.
2. To study the implementation of the dual-intervention into ARV clinics in sub-Saharan African countries while evaluating its effectiveness (HPV vaccination & cervical screening vs cervical screening alone) in reducing HPV infections (and therefore, the risk of cervical precancer and cancer) among WLWH aged 25-35 years.
3. To assess the integration of the dual intervention in HIV clinical services and identify facilitators and barriers for the sustainability of proven effective interventions (dual-intervention, HPV cervical screening) in SSA.

H2VICTORY will include WLWH aged 25-35 years attending ARV clinics to complete HPV vaccination schemes (0-2-6-month) and to be screened with HPV testing. Participants will be evenly allocated (1:1:1) to receive HPV vaccine (3-doses or 1-dose) or placebo. WLWH in a single-dose HPV vaccination scheme will receive placebo at months 2 and 6. Follow-up visits would be scheduled at i) 2 and 6 months to complete vaccination schemes, ii) 12 months 12 (only HPV positives at screening) to complete HPV-based cervical screening according to WHO guidelines, and iii) at 24 months (all participants) to measure efficacy outcomes. Ablative treatment would be offered to those who test positive on HPV at entry and/or at 12 months according to WHO cervical cancer screening and treatment guidelines to progressively remove HPV infections present at baseline. Ablative treatment will be thermal ablation (TA) or cryotherapy (whichever is available) for eligible women (i.e., visualization of the transformation zone and no suspicion of cervical cancer). Women not eligible for TA/cryotherapy would be referred to colposcopy to assess the type of treatment (e.g., LLETZ).

Cervical samples for HPV testing and genotyping will be collected at entry, 12 months (for HPV positives at entry), and 24 months (for everyone), and blood samples for neutralizing HPV antibodies detection will be collected at entry and 24 months (for everyone). The study will initially start in four study centers in South Africa (Cape Town and Durban), Kenya (Nairobi), and Eswatini (Mbabane) where at least 500 participants will be included in each center. HPV vaccine available in school-based programs in each country will be used (i.e., bivalent in South Africa, quadrivalent in Kenya and Eswatini). Hepatitis A (HAV) vaccine will be administrated as a placebo. An experienced pharmacist will be in charge of preparing jabs according to randomization. Central computed randomization will be done. An experienced pharmacist will prepare identical appearance jabs with HPV vaccine or HAV vaccine according to assignation. Allocation will be blinded for participants, care providers, statisticians, and any other staff members. Permuted blocks size 3, and 6 will be used. Additional study centers and collaborators will be involved to extend the study to other countries and settings in order to reach the sample size.

ELIGIBILITY:
Inclusion Criteria:

* Women living with HIV (WLWH)
* Aged 25-35 years
* Attending ARV clinics
* Mentally competent to give informed consent

Exclusion Criteria:

* Pregnancy
* Less than 3 months postpartum
* Women without a cervix (e.g., hysterectomy)
* Plans to move to another city in the next 2 years or any other reason to prevent finalizing the study

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with cervix
Enrollment: 8000 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
HPV infection | 24 months
  HPV prevalent infections at 24 months since initial screening

SECONDARY OUTCOMES:
HPV antibodies | 24 months
  Neutralizing antibodies of HPV at entry and at 24 months
CD4 | 24 months
  CD4 counts at entry and at 24 months
HIV viral load | 24 months
  HIV viral load at entry and at 24 months
Adverse events (AEs) | 24 months
  Adverse events
Serious adverse events (SAEs) | 24 months
  SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Maribel Almonte, MPH, MSc, PhD, Principal Investigator — International Agency for Research on Cancer; Armando Baena, MSc, PhD, Principal Investigator — International Agency for Research on Cancer; Rolando Herrero, MD, PhD, Study Chair — International Agency for Research on Cancer; Mathilde Forestier, PhD, Study Chair — International Agency for Research on Cancer; Joan Valls, MSc, PhD, Study Chair — International Agency for Research on Cancer; Laura Downham, MSc, Study Chair — International Agency for Research on Cancer; Prajakta Adsul, MBBS, MPH, PhD, Study Chair — University of New Mexico; Hennie Botha, MD, PhD, Study Chair — University of Stellenbosch; Haynes van der Merwe, MD, PhD, Study Chair — University of Stellenbosch; Motshedisi Sebitloane, MBChB, PhD, Study Chair — University of KwaZulu; Themba Ginindza, MSc, MPH, PhD, Study Chair — University of KwaZulu; Samah R Sakr, MBChB, Study Chair — Coptic Hope Center; Michael H Chung, MD, MPH, PhD, Study Chair — Emory University; Xolisile Dlamini, MPH, Study Chair — National Cancer Control Unit - Eswatini Ministry of Health; Florence A Anabwani-Richter, MBChB, MPH, Study Chair — Baylor College of Medicine Children's Foundation; Lisbeth Lebelo, PhD, Study Chair — Sefako Makgatho Health Sciences University; Marleen Temmerman, MD, PhD, Study Chair — Aga Khan University; Jean-Marie Dangou, PhD, Study Chair — World Health Organization (AFRO/WHO); Nathalie Broutet, MD, PhD, Study Chair — World Health Organization; Sami L Gottlieb, PhD, Study Chair — World Health Organization; Paul Bloem, MSc, Study Chair — World Health Organization; Soe Soe Thwin, MSc, PhD, Study Chair — World Health Organization; Ajay Rangaraj, MD, MSc, Study Chair — World Health Organization

IPD SHARING:
Plan to Share IPD: Undecided
Plan to be defined